CLINICAL TRIAL: NCT05882487
Title: Safety and Efficacy Study of KL002 in the Treatment of Advanced Primary Parkinson's Dissease
Brief Title: Safety and Efficacy Study of KL002 in the Treatment of Advanced Primary PD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: R&D Kanglin Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0013
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; KL002; Putamen; Stereotactic brain surgery
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KL002 injection solution (Experimental): single dose, neurosurgically infused, bilaterally into the striatum
  Interventions: Genetic: KL002 injection solution

INTERVENTIONS:
Genetic: KL002 injection solution — Neurosurgical delivery of KL002 to the brain

SUMMARY:
This is a non-randomized, open label, dose-escalation study to evaluate the safety and efficacy of KL002 in the treatment of advanced primary Parkinson's disease.

Condition or disease: Parkinson's Disease Intervention/treatment: Drug: KL002 Phase: NA

DETAILED DESCRIPTION:
9 patients will be enrolled to this open-label dose escalation study to evaluate up to three dose levels of KL002 of three patients each. All patients will receive bilateral intraputaminal injections of KL002 through stereotactic brain surgery. The safety and potential clinical responses to KL002 will be assessed by clinical evaluations of Parkinson's disease, cognitive tests, laboratory blood tests and neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

1. Males/females between 40 and 70 years (inclusive)
2. Diagnosed with idiopathic Parkinson's disease, Hoehn and Yahr stage 4 and 5
3. Disease duration at least 5 years
4. MDS UPDRS Part III (total motor) score ≥ 25 and a maximum of 60 in the OFF state
5. Good compliance and can complete all follow-up in accordance with the protocol requirements

Exclusion Criteria:

1. Prior brain surgery including deep brain stimulation or abnormal brain imaging.
2. Presence of depression as measured by Hamilton Depression Scale ≥20
3. History of brain injury or central nervous system infection.
4. Cognitive impairment score<26 on MoCA and ≤ 20 on MMSE dementia scale
5. Evidence of significant medical or psychosis, such as dementia, psychosis, and a history of drug abuse
6. Atypical or secondary parkinsonism, including but not limited to symptoms believed to be due to trauma, brain tumor, infection, cerebrovascular disease, other neurological disease, or to drugs, chemicals, or toxins.
7. Prior gene therapy.
8. Chronic immunosuppressive therapy, including chronic steroids, immunotherapy, cytotoxic therapy and chemotherapy
9. Any other conditions that the investigator believed unsuitable for participation in this study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Day 0 through month 24
  Safety and Tolerability of KL002 assessed by Treatment Emergent Adverse Events

SECONDARY OUTCOMES:
Parkinson's Symptoms | Day 0 through month 24
  Effect of KL002 on Parkinson's symptoms as recorded in subject diaries, neurological, motor, and non-motor assessments, quality of life surveys and changes to Parkinson's medications.
PET Scan Imaging | Day 0 through month 24
  Relationship between KL002 distribution in the brain and change in dopamine expression as indicated in PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Baorong Zhang, M.D., Principal Investigator — The Second Affiliated Hospital Zhejiang University School of Medicine Hangzhou, Zhejiang province, China, 310009
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No